CLINICAL TRIAL: NCT01923779
Title: An Optional Follow-Up Study to Evaluate the Continued Efficacy of ToleroMune Grass in Grass Allergic Subjects Following Challenge With Grass Allergen in an Environmental Exposure Unit
Brief Title: ToleroMune Grass Follow on Study
Status: Completed | Type: Observational
Sponsor: Circassia Limited (Industry)
Collaborators: Adiga Life Sciences, Inc. (Industry); Pharm-Olam International (Industry)
Responsible Party: Sponsor
Other Study IDs: TG002a
Record Dates: First submitted 2013-07-16; First posted 2013-08-16 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Grass Allergy; Rhinoconjunctivitis
Keywords: Grass allergy; Rhinoconjunctivitis; Environmental Exposure Unit; Immunotherapy; ToleroMune Grass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TG002 Subjects: Subjects previously randomised in study TG002

SUMMARY:
Grass pollen allergens are recognised as a major cause of allergic diseases in humans and animals. Worldwide, at least 40% of allergic patients are sensitised to grass pollen allergens and between 50-90% of hayfever or seasonal allergy sufferers are allergic to grass pollen. ToleroMune Grass is a novel, synthetic, allergen-derived peptide desensitising vaccine, currently being developed for the treatment of grass allergy.

The purpose of this optional observational follow-on study is to further evaluate rhinoconjunctivitis symptoms on exposure to Grass in the EEU among subjects who completed all dosing visits in study TG002 approximately one year after the start of treatment.

DETAILED DESCRIPTION:
Subjects who completed all dosing visits and the post treatment challenge (PTC) in study TG002 will be invited to attend the Screening Visit for TG002a. Subjects will attend for 4 visits to the EEU on successive days. Following the last EEC visit a follow-up visit will be performed 3-10 days later.

ELIGIBILITY:
Inclusion Criteria:

* Previously randomised into study TG002, completed all treatment visits and PTC during calendar year 2012.

Exclusion Criteria:

* "Partly controlled" and "uncontrolled" asthma
* History of anaphylaxis to grass allergen
* FEV1 <80% of predicted.
* Treatment with beta-blockers, alpha-adrenoreceptor blockers, tranquilizers or psychoactive drugs
* Symptoms of a clinically relevant illness
* Subjects who cannot tolerate allergen challenge in the EEC

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject previously randomised in study TG002 and completed all dosing visits and the PTC
Sampling Method: Non-Probability Sample
Enrollment: 163 (Estimated)
Dates: Start 2013-05; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Total Rhinoconjunctivitis Symptom Score | Eighteen months post first dose in TG002

SECONDARY OUTCOMES:
Symptom scores for nasal and non nasal symptoms | Eighteen months post first dose in TG002
Skin prick wheal diameter | Eighteen months post first dose in TG002
Peak Nasal Inspiratory Flow | Eighteen months post first dose in TG002
Grass specific IgA | Eighteen months post first dose in TG002
Grass specific IgE | Eighteen months post first dose in TG002
Grass specific IgG4 | Eighteen months post first dose in TG002
Adverse Events | Eighteen months post first dose in TG002

REFERENCES:
- [Derived] Ellis AK, Frankish CW, Armstrong K, Steacy L, Tenn MW, Pawsey S, Hafner RP. Persistence of the clinical effect of grass allergen peptide immunotherapy after the second and third grass pollen seasons. J Allergy Clin Immunol. 2020 Feb;145(2):610-618.e9. doi: 10.1016/j.jaci.2019.09.010. Epub 2019 Sep 27. PMID 31568796